CLINICAL TRIAL: NCT05853172
Title: Surgical Conversion of Candonilimab (AK104) Combined With Paclitaxel, S-1 and Apatinib for Unresectable Advanced Gastric(G)/Gastroesophageal Junction(GEJ) Cancer
Brief Title: Surgical Conversion of Candonilimab (AK104) Plus Paclitaxel, S-1 and Apatinib for Unresectable Advanced G/GEJ Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20221047
Record Dates: First submitted 2023-04-24; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 plus apatinib, paclitaxel and S-1 (Experimental): AK104 (10mg/kg, iv, Q3W) is combined with apatinib (250mg, po, qd), paclitaxel (non-peritoneal metastasis: 130mg/m2, iv, D1; peritoneal metastasis: 90mg/m2, iv, 40mg/m2, ip, D1) and S-1(60mg, po, bid, D1-D14) for up to 6 cycle for up to 6 cycles.
  Interventions: Drug: AK104; Drug: Apatinib; Drug: Paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: AK104 — Subjects will receive AK104 until disease progression or for up to 6 cycles.
Drug: Apatinib — Subjects will receive apatinib until disease progression or for up to 6 cycles.
Drug: Paclitaxel — Subjects will receive paclitaxel until disease progression or for up to 6 cycles.
Drug: S-1 — Subjects will receive S-1 until disease progression or for up to 6 cycles.

SUMMARY:
This is a prospective, single-arm, open-label，single-center, phase II study, aiming to to evaluate the surgical conversion feasibility of AK104 combined with apatinib, paclitaxel and S-1 in unresectable stage IV G/GEJ cancer.

DETAILED DESCRIPTION:
Eligible patients receive AK104 (10mg/kg, iv, Q3W) combined with apatinib (250mg, po, qd), paclitaxel (non-peritoneal metastasis: 130mg/m2, iv, D1; peritoneal metastasis :90mg/m2, iv, 40mg/m2, ip, D1) and S-1(60mg, po, bid, D1-D14) for up to 6 cycles. Patients assessed by Multi-Disciplinary Treatment (MDT) to meet the criteria for surgical resection undergo gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
2. Clinically diagnosed unresectable stage IV gastric (G) or gastroesophageal junction (GEJ) adenocarcinoma by CT/MRI/Positron Emission Tomography (PET) -CT.
3. Not received prior systemic therapy for stage IV G/GEJ adenocarcinoma
4. At least one measurable tumor lesion per RECIST v1.1;
5. Major organ functions are adequate;
6. Expected survival is ≥ 3 months;
7. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1;

Exclusion Criteria:

1. Human Epidermal GrowthFactor Receptor 2 (HER2)-positive G/GEJ adenocarcinoma;
2. Previously received immune checkpoint inhibitors, including but not limited to programmed death 1 (PD-1) inhibitors and cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors;
3. Central nervous system, lung, or bone metastases;
4. Known history of active or autoimmune disease;
5. Known history of other malignancies;
6. Known history of severe cardiovascular and cerebrovascular diseases;
7. Known history of gastrointestinal bleeding within the past 3 months or significant tendency to gastrointestinal bleeding;
8. Active infection or fever of unknown origin;
9. Known history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severe impairment of lung function;
10. Known history of immunodeficiency, positive HIV antibody (HIVAb) test, or other acquired or congenital immunodeficiency disorder, or active hepatitis;
11. Known history of mental disorder or psychoactive substance abuse;
12. Hypersensitivity to the drugs of this regimen;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
R0 surgical conversion rate | up to 2 years

SECONDARY OUTCOMES:
R0 resection rate | up to 2 years
Pathological complete response (pCR) | up to 2 years
Pathological major response (MPR) | up to 2 years
Objective response rate (ORR) | up to 2 years
Disease control rate (DCR) | up to 2 years
Progression-free survival (PFS) | up to 2 years
Adverse event (AE) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No